CLINICAL TRIAL: NCT07305233
Title: The Effect of Web-Supported Interactive Learning on the Knowledge Level of Nursing Students on Pediatric Drug Dose Calculation: A Randomized Controlled Study
Brief Title: Pediatric Drug Dose Calculation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Dilek Zengin, Assisstant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 741023
Record Dates: First submitted 2025-11-26; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Drug Dose
Keywords: Pediatric nursing; drug calculation; ınteractive learning

STUDY DESIGN:
Intervention Model Description: Third-year nursing students take the Diseases and Nursing Care II lecture in the autumn term. Students do 1 week of laboratory practice after 3 weeks of theoretical course education. In laboratory practice, they receive training on Pediatric Drug Dose Calculation. Before starting the laboratory practice for the project study, a face-to-face meeting was planned before the major courses were attended by all 3rd year students and students were informed about the purpose, goal, and procedures of the study. The students were informed that participation in the study was voluntary and would not affect their academic achievement in any way. The first 108 students who were willing to participate in the study were included in the study and were assigned to the control and study groups according to the randomization list. Data collection for both groups was carried out as follows.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control Group (n=54) Day 1 The aim, objective, and study steps of the study were verbally explained to participants in a face-to-face meeting. The students were informed that they could withdraw from the study for any reason at any stage of the study and that their participation in the study would not affect their academic achievement. In addition, students' written consent was obtained through the voluntary consent form containing all these statements. The students were placed according to the exam order and were first asked to fill in the "Individual Identification Form". Once all the students completed the form, they were informed about the content and duration of the "Drug Dose Calculation Knowledge Test" pretest, which they then completed within 30 minutes.
  Day 2 Face-to-face training was given to the students in this group via a "Pediatric Drug Dose Calculation" PowerPoint presentation. The training was supported with visual materials and active participation of students was ens
- study group (Experimental): Study Group (n=54):
  Day 1 The aim, objective, and study steps of the study were verbally explained to participants in a face-to-face meeting. The students were informed that they could withdraw from the study for any reason at any stage of the study and that their participation in the study would not affect their academic achievement. In addition, students' written consent was obtained through the voluntary consent form containing all these statements. The students were placed according to the exam order and were first asked to fill in the 'Individual Identification Form'. Once all the students completed the form, they were informed about the content and duration of the 'Drug Dose Calculation Knowledge Test' pretest, which they then completed within 30 minutes.
  Day 2 Face-to-face training was given to the students in this group via a "Pediatric Drug Dose Calculation" PowerPoint presentation. The training was supported with visual materials and active participation of the students was
  Interventions: Other: Study Group

INTERVENTIONS:
Other: Study Group — The study was conducted with nursing students who were verbally informed about the aim, objectives, and procedures in a face-to-face meeting. They were told that participation was voluntary, could be withdrawn at any time, and would not affect academic performance. Written consent was obtained. On Day 1, students filled in the "Individual Identification Form" and completed the "Drug Dose Calculation Knowledge Test" pretest within 30 minutes. On Day 2, face-to-face training on "Pediatric Drug Dose Calculation" was provided using a PowerPoint presentation supported by visuals and interactive discussions. Students were then introduced to an interactive Edpuzzle application, informed about its use, access, and feedback features, and allowed to use it anytime. On Day 9, one week later, the post-test of the knowledge test was administered, followed by the "Perceived Learning Scale" and "Medication Administration Self-Efficacy Scale in Children for Nursing Students."
  Arms: study group

SUMMARY:
This study is a randomized controlled trial that aimed to investigate the effect of a web-supported interactive learning program on the knowledge level of nursing students about pediatric drug dose calculation.

The study was conducted at one of Turkey's most established nursing faculties, and 108 students participated in the study. Participants were randomly assigned to study (n:54) and control (n:54) groups. The study group received both a traditional lecture and a Web-supported interactive learning application, while the control group was limited to a traditional lecture-based instruction. The "Drug Dose Calculation Knowledge Test", "Perceived Learning Scale", and "Medication Administration Self-Efficacy Scale in Children for Nursing Students" scales were used to collect the data.

DETAILED DESCRIPTION:
Purpose and Type of Research This study aimed to investigate the effect of a web-supported interactive learning program on the knowledge level of nursing students about pediatric drug dose calculation. This randomized controlled trial with two parallel groups (pretest and posttest design) was conducted in accordance with the Consolidated Standards of Reporting Trials (CONSORT) checklist.

Population and Sample of the Study This study was conducted at a Nursing Faculty located in Western Turkey. The population of this study consisted of 3rd-year students (n = 346) studying at the Faculty of Nursing for the first time in the first semester of the 2022-2023 academic year. The research sample was determined through a power analysis using the G*Power 3.1.9.2 program under the Repeated Measures ANOVA test to identify the significant difference between the groups before and after the training. For the analysis, with an alpha level of 0.05, an effect size of 0.25, and 80% power, a minimum sample of 98 (49 people per group) was found sufficient. To account for potential data loss in the sample group, a total of 108 students -10% more than the sample number- were included in the study. A simple randomization method was used for sample selection and a randomization list was determined. The participants were assigned to the study and control groups according to the randomization list.

Third-year undergraduate nursing students enrolled in the Diseases and Nursing Care II lecture for the first time in the first semester of the 2022-2023 academic year were invited to participate in this study. Students who had a computer or smartphone and students who volunteered to participate in the study were included in the study. Students who did not have a computer or smartphone and students who did not complete all stages of the study were excluded from the study.

Data Collection and Analysis Third-year nursing students take the Diseases and Nursing Care II lecture in the autumn term. Students do 1 week of laboratory practice after 3 weeks of theoretical course education. In laboratory practice, they receive training on Pediatric Drug Dose Calculation. Before starting the laboratory practice for the project study, a face-to-face meeting was planned before the major courses were attended by all 3rd year students and students were informed about the purpose, goal, and procedures of the study. The students were informed that participation in the study was voluntary and would not affect their academic achievement in any way. The first 108 students who were willing to participate in the study were included in the study and were assigned to the control and study groups according to the randomization list. Data collection for both groups was carried out as follows.

Control Group (n=54) Day 1 The aim, objective, and study steps of the study were verbally explained to participants in a face-to-face meeting. The students were informed that they could withdraw from the study for any reason at any stage of the study and that their participation in the study would not affect their academic achievement. In addition, students' written consent was obtained through the voluntary consent form containing all these statements. The students were placed according to the exam order and were first asked to fill in the "Individual Identification Form". Once all the students completed the form, they were informed about the content and duration of the "Drug Dose Calculation Knowledge Test" pretest, which they then completed within 30 minutes.

Day 2 Face-to-face training was given to the students in this group via a "Pediatric Drug Dose Calculation" PowerPoint presentation. The training was supported with visual materials and active participation of students was ensured with question-answer interactions.

Day 9 One week after the training, the "Drug Dose Calculation Knowledge Test" post-test was applied, with students seated according to their exam order. Students were given 30 minutes to complete the post-test. After completing the post-test, the "Perceived Learning Scale", which enables the student to make a self-assessment on the subject, and the "Medication Administration Self-Efficacy Scale in Children for Nursing Students", which enables the student to make a self-assessment on drug administration, were distributed and the scales were filled in.

Study Group (n=54):

Day 1 The aim, objective, and study steps of the study were verbally explained to participants in a face-to-face meeting. The students were informed that they could withdraw from the study for any reason at any stage of the study and that their participation in the study would not affect their academic achievement. In addition, students' written consent was obtained through the voluntary consent form containing all these statements. The students were placed according to the exam order and were first asked to fill in the 'Individual Identification Form'. Once all the students completed the form, they were informed about the content and duration of the 'Drug Dose Calculation Knowledge Test' pretest, which they then completed within 30 minutes.

Day 2 Face-to-face training was given to the students in this group via a "Pediatric Drug Dose Calculation" PowerPoint presentation. The training was supported with visual materials and active participation of the students was ensured with question-answer interactions. After the verbal training was completed, the students were informed about the use of the interactive learning application created through the Edpuzzle program. Information was given about how to access the application, how to answer the questions in the interactive application, how to use the Edpuzzle application, and how students can see the correct and incorrect applications in the interactive video. Students were also informed that they could access the interactive application at any time, from any location, and as often as they desired.

Day 9 One week after the training, the "Drug Dose Calculation Knowledge Test" post-test was applied, with students seated according to their exam order. Students were given 30 minutes to complete the post-test. After completing the post-test, the "Perceived Learning Scale", which enables the student to make a self-assessment on the subject, and the "Medication Administration Self-Efficacy Scale in Children for Nursing Students", which enables the student to make a self-assessment on drug administration, were distributed and the scales were filled in.

Data Collection Instruments The study data were collected using the 'Individual Identification Form', "Drug Dose Calculation Knowledge Test", "Perceived Learning Scale" and "Medication Adminstration Self-Efficacy Scale in Children for Nursing Students".

Individual Identification Form: The form, developed by the researchers, consisted of 5 questions including age, gender, graduated school, achievement status, and satisfaction with the nursing profession.

Drug Dose Calculations Knowledge Test: It was prepared by the researchers in line with the relevant literature. Each item in the test has a different scoring scheme. The Pediatric Drug Dose Calculations Knowledge Test consists of a total of 17 items including 6 conversion calculations, 3 safe dose range calculations, 1 drug dose calculation, 5 calculations including dry powder volume, 1 body surface area calculation formula, and 1 definition of dry powder volume. Expert opinion was taken for the content validity of the test.

Perceived Learning Scale: The Turkish validity and reliability of the scale was established. Consisting of 9 items, the scale has three factors to measure cognitive, affective, and psychomotor perceived learning. The total score of the scale varies between 9-63 and it takes 3-5 minutes to complete the scale. The Cronbach's Alpha reliability coefficient of the scale is 0.79. Permission was obtained from the authors for the use of the scale.

Medication Administration Self-Efficacy Scale in Children for Nursing Students: The scale aims to determine the self-efficacy levels of nursing students regarding drug administration in children. It consists of 16 items and 2 sub-scales. Total scores range from 16 to 80, with higher scores indicating greater self-efficacy in pediatric drug administration. The Cronbach's alpha coefficient was 0.94for the overall scale, 0.91 for the first drug preparation sub-scale, and 0.87 for the second drug administration sub-scale. Permission was obtained from the authors for the use of the scale.

Pediatric Drug Dose Calculation PowerPoint Presentation: The presentation was prepared by the project team based the relevant and current literature. Pediatric Drug Dose Calculation PowerPoint presentation includes the responsibility of the pediatric nurse in drug administration, how drug dose calculation is performed in pediatrics, determination of the safe dose range of drugs, dry powder volume, conversion calculations and drug calculation examples.

Pediatric Drug Dose Calculation Interactive Application: The interactive application is a video game prepared in line with the relevant literature to include the responsibility of the pediatric nurse in drug administration, how drug dose calculation is performed in pediatrics, determination of the safe dose range of drugs, dry powder volume, conversion calculations and drug calculation examples. The video content was prepared to be the same as the PowerPoint presentation. After the filming was completed by the researchers, the videos were edited by the experienced researcher. During the video shooting, pediatric drug dose calculation was mentioned comprehensively to make students aware of their mistakes and to minimize the risk of dose error. To edit the video content, the video was uploaded to the Edpuzzle program by logging in as an educator. Open-ended and multiple-choice questions that students should answer in the video were embedded in the 'edit' section in the 'Video Preview' section of the Edpuzzle application. A team was created via the Microsoft Teams application for students to access the edited video content. A class was assigned to the team created with Microsoft Teams from Eddpuzzle, which allowed tracking of correct and incorrect responses by students.

ELIGIBILITY:
Inclusion Criteria:

Students who had a computer or smartphone and students who volunteered to participate in the study were included in the study

Exclusion Criteria:

Students who did not have a computer or smartphone and students who did not complete all stages of the study were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
knowledge level | 9 days
  Knowledge level of nursing students about pediatric drug dose calculation by using the Drug Dose Calculation Knowledge Test. The Pediatric Drug Dose Calculations Knowledge Test consists of a total of 17 items including 6 conversion calculations, 3 safe dose range calculations, 1 drug dose calculation, 5 calculations including dry powder volume, 1 body surface area calculation formula, and 1 definition of dry powder volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I have not decided yet.